CLINICAL TRIAL: NCT05113121
Title: Correlation Between Pupil Size and Ocular Signs in Pseudoexfoliation Syndrome (PEX): a Contralateral Eye Study.
Brief Title: Correlation Between Pupil Size and Ocular Signs of Pseudoexfoliation Syndrome
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud F. Rateb, Associate Professor, Assiut University
Other Study IDs: PEXPUPIL
Record Dates: First submitted 2021-10-28; First posted 2021-11-09 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Pseudoexfoliation Syndrome; Pseudoexfoliation Glaucoma in Both Eyes; Pseudoexfoliation of Lens; Glaucoma
Keywords: cataract; glaucoma
MeSH Terms: conditions — Exfoliation Syndrome; Glaucoma; Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: , Humphrey visual field (24-2) analysis and optical coherence tomography on retinal nerve fiber layer (RNFL) and ganglion cell complex.(GCC) — , Humphrey visual field (24-2) analysis and optical coherence tomography on retinal nerve fiber layer (RNFL) and ganglion cell complex.(GCC)

SUMMARY:
To study possible correlation between the size of the pupil in both room light and after dilation between both eyes in bilateral pseudoexfoliation with Intraocular pressure, lens clarity and stability, Optic disc , Visual changes and glaucoma changes by optical coherence tomography

DETAILED DESCRIPTION:
For each patient. Full preoperative ophthalmological assessment will be done using slit lamp , size of the pupil in regular room light (usually around 2000 Lux) and post dilation with tropicamide 1%. baseline IOP measurement using Goldmann applanation tonometer, UCDVA (Uncorrected Distance Visual Acuity)and CDVA (Corrected Distance visual acuity), lens opacification or clarity, stability or subluxation. corneal endothelial cell count. Fundus examination using 90 D or 78D lenses, Humphrey visual field (24-2) analysis and optical coherence tomography on retinal nerve fiber layer (RNFL) and ganglion cell complex.(GCC)

ELIGIBILITY:
Inclusion Criteria:

All patients with pseudoexfoliation syndrome

Exclusion Criteria:

previous ocular surgery or ocular trauma affecting pupil. Any systemic or neurologic disease affecting pupil

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients , age : 18 years and older
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
correlation between pupil size and severity of Pseudoexfoliation | 2-3 months
  in each eye of the same patient we study correlation between pupil size with ntraocular pressure, lens status, corneal endothelial count and glaucomatous damage represented by (optic disc changes (cup to disc ratio) and OCT changes (RNFL and GCC)

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Rateb, Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
IPD can be shared upon request after completion of the research
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after completion of data and for five years.
Access Criteria: It will be upon request through email

REFERENCES:
- [Background] Shazly TA, Farrag AN, Kamel A, Al-Hussaini AK. Prevalence of pseudoexfoliation syndrome and pseudoexfoliation glaucoma in Upper Egypt. BMC Ophthalmol. 2011 Jun 27;11:18. doi: 10.1186/1471-2415-11-18. PMID 21707986
- [Background] Plateroti P, Plateroti AM, Abdolrahimzadeh S, Scuderi G. Pseudoexfoliation Syndrome and Pseudoexfoliation Glaucoma: A Review of the Literature with Updates on Surgical Management. J Ophthalmol. 2015;2015:370371. doi: 10.1155/2015/370371. Epub 2015 Oct 29. PMID 26605078
- [Background] Tekin K, Kiziltoprak H, Sekeroglu MA, Yetkin E, Bayraktar S, Yilmazbas P. Static and dynamic pupil characteristics in pseudoexfoliation syndrome and glaucoma. Clin Exp Optom. 2020 May;103(3):332-338. doi: 10.1111/cxo.12945. Epub 2019 Jul 30. PMID 31364197
- [Background] Akman A, Yilmaz G, Oto S, Akova YA. Comparison of various pupil dilatation methods for phacoemulsification in eyes with a small pupil secondary to pseudoexfoliation. Ophthalmology. 2004 Sep;111(9):1693-8. doi: 10.1016/j.ophtha.2004.02.008. PMID 15350324